CLINICAL TRIAL: NCT03905681
Title: The Use of Transcutaneous Electrical Nerve Stimulation on the Efficacy of Acute Back Pain Within an Emergency Department Triage: A Randomized Trial
Brief Title: TENS Efficacy on Acute Back Pain in an Emergency Department Triage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Beaumont Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Manley, Captain David Manley, PA-C, Emergency Medicine Physician Assistant Resident, William Beaumont Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.2019.027d
Record Dates: First submitted 2019-03-30; First posted 2019-04-05 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Acute Back Injury
Keywords: Transcutaneous Electrical Nerve Stimulation, Acute back pain
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Using a sample population in a military treatment facility emergency department, this prospective, randomized controlled trial utilized forty-six total participants evenly divided to both a active and placebo group, were used to determine the efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) on acute back pain of ambulatory patients presenting for emergent care.
Who Masked: Participant, Care Provider
Masking Description: After computer-generated randomization, participants will either receive the active TENS treatment for 30 minutes, or receive the application of TENS pads and wear the device with no electrical stimulation. Both groups will have pre and post visual analogue scores assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TENS Group "Group A" (Active Comparator): After all necessary data collection forms are obtained, a pre-VAS score will be obtained. The participant will point to the area of maximum subjective pain, and then four TENS pads will be applied directly around the point of maximal pain that was determined by the patient, located at least 3 centimeters but no more than 6 centimeters from the area in a square or frame-like placement. While the device is off, it will be set at the following settings: The selector switch will be set to 'Milli' or milliamperes, and the frequency dial will be rotated to 100 Hertz. The participant will be instructed to rotate both dials in a clockwise direction if more intensity is desired, or counter-clockwise if less intensity is desired. The participant will wear the device and pads for a 30-minute duration; upon completion, post-VAS scores and a patient satisfaction survey will be obtained.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation
- Placebo TENS Group "Group B" (Placebo Comparator): After all necessary data collection forms are obtained, a pre-VAS score will be obtained. The participant will point to the area of maximum subjective pain, and then four TENS pads will be applied directly around the point of maximal pain that was determined by the patient, located at least 3 centimeters but no more than 6 centimeters from the area in a square or frame-like placement. However, no electrical stimulation will be provided. The participant will also wear the device and pads for a 30-minute duration; upon completion, post-VAS scores and a patient satisfaction survey will be obtained.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Application of TENS pads and wearing of the TENS device.
  Other Names: TENS

SUMMARY:
Transcutaneous Electrical Nerve Stimulation (TENS) devices produce a gentle electrical stimulation that when applied through pads applied directly to the skin, has a noticeable effect in reducing pain associated with various types of injuries and ailments. Several recent studies have shown efficacy when used for acute pain specific to primary dysmenorrhea, renal colic, lower-extremity pain, and pain associated with spinal cord injury, and was achieved without adverse effects. This study is intended to compare the effects of TENS units on acute back pain on ambulatory patients who are awaiting emergency medical treatment, to uncover if a statistically-significant analgesic effect is noted compared to a placebo device.

DETAILED DESCRIPTION:
With the emerging amount of new data on the treatment specific to acute pain, it is theorized that early TENS application can be an adjunct for acute pain reduction, specifically for patients awaiting treatment in an emergency department triage waiting room. TENS stimulators are advantageous to patients in that they are non-pharmacologic and non-invasive therapy. TENS devices have an excellent safety profile, are associated with very few contraindications, and have negligible side-effects or adverse events: the most common being minor skin irritation. (Sluka and Walsh 2003) Of financial benefit to a hospital considering their implementation, these devices are also inexpensive. In the realm of emergency medicine, which is being scrutinized to reduce opioid prescriptions, measures must be taken to maximize the efficacy of alternative pain-relief adjuncts.

There are significant gaps in the literature which have depicted no significant benefits compared to physical therapy and other modalities. These studies had used variable treatments times and frequencies, which were not solidified in scientific research at the time of their results. The use of these stimulators has been extensively studied, and the evidence to support their use on various conditions has been inconclusive. Early meta-analyses and systematic reviews have noted the data are inconsistent to suggest a mean reduction of pain when assessed on chronic pain. (Brosseau et al. 2002) However, when applied extensively and at regular settings, TENS has shown the presence of tolerance to TENS when used chronically in as few as four days. (Chandran and Sluka, 2003) This study is intended to harness the newest research comparing the most-effective settings and durations of TENS units, and compare the effects of TENS units on acute back pain on ambulatory patients who are awaiting emergency medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presents to the Emergency Department in an ambulatory status
* Has a complaint of traumatic back pain, acute or acute-on-chronic, which is 3 weeks or less in duration.
* Is designated to an Emergency Severity Index Category of 4 or 5.
* Patient must be unfamiliar with TENS use
* Projected wait time of greater than 30 minutes before a visit with an Emergency Department provider is anticipated based on triage category
* Not actively pregnant for female patients

Exclusion Criteria:

* Patient has a history of using TENS in the past
* Patient is actively pregnant
* History of narcotic use or abuse in the last 24 hours
* Patient has a cardiac pacemaker or a neurostimulation-implant device
* Patient is designated to an Emergency Severity Index Category of 1, 2, or 3
* Patient has an open wound, abrasion, skin rash, or tattoo < 6 weeks old where pads will be placed
* Patient has a current history of Low Back Pain 'red flags' (Bilateral radicular symptoms, saddle anesthesia or paresthesia, bladder incontinence, or bowel incontinence) which require immediate attention.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Decrease in pain using Visual Analogue Scores (VAS) | After 30-minute duration of treatment
  Enrolled participants will have baseline Visual Analogue Scores (VAS) pain scale scores assessed, consisting of a 0 to 100 unit scale, with instruction to locate their level of pain on the scale of 0 being "No pain at all," 50 being "Moderate Pain," and 100 being "Worst pain imaginable," and will be compared to score on the same scale after treatment.

SECONDARY OUTCOMES:
Increase in patient satisfaction while awaiting treatment | After 30-minute duration of treatment
  Using an assessment questionnaire of patient satisfaction, with nominal and ordinal results measured for statistical significance:
  1. Do you feel that early intervention with this device increases your satisfaction as a patient?
  2. If given the opportunity, would you like to continue to use this device while waiting?
  3. If you were to guess, do you think you were part of the treatment group or the no-treatment group?
  4. On a scale of 1 through 10, with 1 being "completely dissatisfied" and 10 being "completely satisfied," how satisfied are you with being provided this treatment?

CONTACTS AND LOCATIONS:
Locations (1):
- William Beaumont Army Medical Center, Fort Bliss, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed, the data used for statistical analysis will be void of personally identifiable information. This data will be in electronic form for use in government-approved software, such as Microsoft Office. These documents will be distributed only to the Primary Investigator and the William Beaumont Army Medical Center (WBAMC) Department of Clinical Investigations assistance with statistical analysis or future publishing consideration. All paper documents are to be maintained in accordance with Department of Clinical Investigations policies; study-specific electronic documents will be kept for a minimum of 3 years before deletion. Upon study closure, all personally identifiable information (including the Master Key) will be destroyed or deleted, and a de-identified data set maintained by the WBAMC Emergency Medicine Physician Assistant Residency Program Director for further study as needed. No human biological specimens will be maintained.
Supporting Information: SAP, ICF
Time Frame: 3 years, or as determined by the WBAMC Department of Clinical Investigations.
Access Criteria: Principal Investigator, WBAMC Department of Clinical Investigations, WBAMC Emergency Medicine Physician Assistant Residency Program Director.

REFERENCES:
- [Background] Bi X, Lv H, Chen BL, Li X, Wang XQ. Effects of transcutaneous electrical nerve stimulation on pain in patients with spinal cord injury: a randomized controlled trial. J Phys Ther Sci. 2015 Jan;27(1):23-5. doi: 10.1589/jpts.27.23. Epub 2015 Jan 9. PMID 25642029
- [Background] Sluka KA, Walsh D. Transcutaneous electrical nerve stimulation: basic science mechanisms and clinical effectiveness. J Pain. 2003 Apr;4(3):109-21. doi: 10.1054/jpai.2003.434. PMID 14622708
- [Background] Brosseau L, Milne S, Robinson V, Marchand S, Shea B, Wells G, Tugwell P. Efficacy of the transcutaneous electrical nerve stimulation for the treatment of chronic low back pain: a meta-analysis. Spine (Phila Pa 1976). 2002 Mar 15;27(6):596-603. doi: 10.1097/00007632-200203150-00007. PMID 11884907
- [Background] Chandran P, Sluka KA. Development of opioid tolerance with repeated transcutaneous electrical nerve stimulation administration. Pain. 2003 Mar;102(1-2):195-201. doi: 10.1016/s0304-3959(02)00381-0. PMID 12620611
- [Background] Lauretti GR, Oliveira R, Parada F, Mattos AL. The New Portable Transcutaneous Electrical Nerve Stimulation Device Was Efficacious in the Control of Primary Dysmenorrhea Cramp Pain. Neuromodulation. 2015 Aug;18(6):522-6; discussion 522-7. doi: 10.1111/ner.12269. Epub 2015 Feb 5. PMID 25655828
- [Background] Ayyildiz A, Akgul T, Nuhoglu B. Re: Transcutaneous electrical nerve stimulation: an effective treatment for pain caused by renal colic in emergency care. B. Mora, E. Giorni, M. Dobrovits, R. Barker, T. Lang, C. Gore and A. Kober, J Urol 2006; 175: 1737. J Urol. 2007 Jan;177(1):405. doi: 10.1016/j.juro.2006.09.013. No abstract available. PMID 17162100
- [Background] Gozani SN. Fixed-site high-frequency transcutaneous electrical nerve stimulation for treatment of chronic low back and lower extremity pain. J Pain Res. 2016 Jun 28;9:469-79. doi: 10.2147/JPR.S111035. eCollection 2016. PMID 27418854